CLINICAL TRIAL: NCT06947733
Title: Analysis of the Effect of Pre-course Videos on Improving Clinical Skills in Emergency Ultrasound Training
Acronym: CVC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Po-Hsiang Liao, Doctor, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024 - 06 - 006B
Record Dates: First submitted 2024-08-08; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Medical Education
Keywords: Point-of-Care Ultrasound

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: subjects randomly assigned to one of three groups: the first-person perspective video group, the face-to-face perspective video group, and the control group (who will not watch any videos).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the first-person perspective video group (Active Comparator): Students will watch first-person point-of-view (POV) filmed videos and will complete both pre- and post-tests on the day of the course.
  Interventions: Behavioral: pre-class videos
- the face-to-face perspective video group (Active Comparator): Students will watch the face-to-face perspective filmed videos and will complete both pre- and post-tests on the day of the course.
  Interventions: Behavioral: pre-class videos
- the control group (who will not watch any videos) (Placebo Comparator): A control group without video viewing will also complete both pre- and post-tests on the day of the course.
  Interventions: Behavioral: no pre-class videos

INTERVENTIONS:
Behavioral: pre-class videos — This project aims to evaluate the impact of pre-class videos on enhancing ultrasound teaching effectiveness, particularly comparing videos shot with a first-person perspective (POV) to those shot with a face-to-face perspective.
  Arms: the face-to-face perspective video group; the first-person perspective video group
Behavioral: no pre-class videos — the control group (who will not watch any videos)
  Arms: the control group (who will not watch any videos)

SUMMARY:
Project Background Point-of-Care Ultrasound (POCUS) has become an important part of medical education in recent years. However, due to limited resources of ultrasound machines and clinical instructors, hands-on practice opportunities are limited, affecting the quality of teaching. Effectively imparting ultrasound operation skills has become a major challenge in improving training quality. This project aims to evaluate the impact of pre-class videos on enhancing ultrasound teaching effectiveness, particularly comparing videos shot with a first-person perspective (POV) to those shot with a face-to-face perspective.

Project Objectives Primary Objective: To evaluate the impact of learning from pre-class videos on enhancing the effectiveness of ultrasound teaching.

Secondary Objective: To investigate the effect of different filming techniques (POV versus face-to-face) on learning outcomes.

Research Design The study will adopt a parallel research design, with subjects randomly assigned to one of three groups: the first-person perspective video group, the face-to-face perspective video group, and the control group (who will not watch any videos).

Procedure on the Day of Instruction Complete a basic information and learning experience questionnaire. Conduct a pre-test practical, recording the operation of the ultrasound. Provide one-on-one instruction, offering detailed operational guidance. Conduct a post-test practical, allowing students to independently perform ultrasound-guided central venous catheter insertion.

Complete a post-test questionnaire. Expected Outcomes This study anticipates that learning through pre-class videos will effectively enhance students' ultrasound operation skills and improve teaching quality. Teaching videos shot with a POV may provide a more realistic learning experience, thereby enhancing students' learning outcomes. By comparing different filming techniques, this project will provide empirical data that can inform future ultrasound teaching methods, ultimately improving the overall effectiveness of medical education.

DETAILED DESCRIPTION:
Study Population Participants included PGY physicians at the hospital, the majority of whom had not previously performed independent CVC insertion or used ultrasound guidance. A total of 72 PGY physicians voluntarily enrolled in the study after receiving invitations via email and posters. No adverse events were reported during the study.

Video Preparation

Instructional videos were recorded in two formats:

First-person POV video using a GoPro mounted on the instructor's head.

Face-to-face (FtF) side-view video using two strategically placed cameras to capture side and front views simultaneously.

Both videos were standardized to 25 minutes and 42 seconds in duration and were uploaded privately on YouTube. Access was restricted to registered participant emails and granted three days prior to training. A cartoon character inserted at the end of each video served as a verification checkpoint during pre-class surveys.

Interventions

Participants were randomized into one of three groups using a block randomization method:

POV first-person video group

Face-to-face side-view video group

Control group (no video)

All participants received a pre-class email. The video groups received access to their assigned instructional video and the CVC checklist, while the control group received only the checklist.

Training Day Procedure

Participants first completed a pre-training questionnaire assessing demographics, procedural experience, and video viewing compliance. This was followed by:

Pre-training assessment: Participants performed ultrasound-guided CVC on a phantom model, evaluated by a competency checklist and global rating score.

One-on-one instruction: Instructors provided standardized guidance.

Post-training assessment: Participants repeated the CVC procedure independently and were re-evaluated.

Post-training questionnaire: Included self-assessed confidence and satisfaction scores.

All assessments were performed by a single instructor who was blinded to group allocation.

Statistical Analysis

Continuous variables were reported as medians with interquartile ranges, and categorical variables as counts and percentages. Normality was assessed, and non-parametric tests were used due to skewed data. Between-group comparisons were performed using:

Kruskal-Wallis test (three-group comparison)

Mann-Whitney U test (two-group comparison)

Wilcoxon signed-rank test (paired pre/post comparison)

Chi-square or Fisher's exact test was used for categorical data. A significance threshold of α = 0.05 was used, with Bonferroni correction applied (adjusted α = 0.0167). Analyses were conducted in Python (version 3.13).

ELIGIBILITY:
Inclusion Criteria:

* PGY physicians
* Medical students

Exclusion Criteria:

* who refused the invitation of this learning project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Checklist Completion Score (0-34 points) | 6 months
  Objective evaluation of procedural steps during central venous catheterization, assessed using a standardized skills checklist.
Global Rating Score (1-10 scale) | 6 months
  Instructor-assigned score reflecting overall procedural fluency and technical competence.

SECONDARY OUTCOMES:
Procedural Time (minutes) | 6 months
  Total time taken to complete the procedure during pre- and post-training assessments. Comparisons will be made between: Participants who received pre-class videos vs. those who did not (pre-test comparison)

CONTACTS AND LOCATIONS:
Overall Officials: Po-Hsiang Liao, MD, Principal Investigator — Department of Emergency Medicine, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
However, researchers interested in accessing de-identified data related to this study can contact us via email after the paper is published. We will consider requests on a case-by-case basis.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT06947733/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT06947733/ICF_001.pdf